CLINICAL TRIAL: NCT04073446
Title: Focal Pain Outcomes Using Configurations Applied for Lateral Stimulation
Acronym: FOCAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A4068
Record Dates: First submitted 2019-07-23; First posted 2019-08-29 (Actual); Results first posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2022-12

CONDITIONS: Chronic Pain
Keywords: Spinal Cord Stimulation; Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Dorsal Column (DC) Perception (Active Comparator): Use of DC Perception based programming
  Interventions: Device: Spinal Cord Stimulation
- Dorsal Root (DR) Perception (Active Comparator): Use of DR Perception based programming
  Interventions: Device: Spinal Cord Stimulation
- Dorsal Root (DR) Sub-perception (Active Comparator): Use of DR sub-perception based programming
  Interventions: Device: Spinal Cord Stimulation
- Dorsal Column (DC) Sub-perception (Active Comparator): Use of DC sub-perception based programming
  Interventions: Device: Spinal Cord Stimulation

INTERVENTIONS:
Device: Spinal Cord Stimulation — Patients eligible for SCS

SUMMARY:
To evaluate programming modalities at various targets for focal foot, knee pain, and groin pain relief.

ELIGIBILITY:
Key Inclusion Criteria:

* Average unilateral foot, or knee or groin pain intensity of 6 or greater on a 0-10 numerical rating scale at Baseline Visit based on 7-day average NRS score
* Subject signed a valid, EC-approved informed consent form (ICF)
* Willing and able to comply with all protocol-required procedures and assessments/evaluations
* 18 years of age or older when written informed consent is obtained

Key Exclusion Criteria:

* Significant cognitive impairment at Screening that, in the opinion of the Investigator, would reasonably be expected to impair the study candidates to participate in the study
* Participating (or intends to participate) in another drug or device clinical trial that may influence the data that will be collected for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roshini Jain, Study Director — Boston Scientific Corporation
Locations (1):
- AZ Nikolaas, Sint-Niklaas, Belgium

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 subjects were enrolled. However 2 were implanted and proceeded to crossover phase
Groups:
- Subjects Received All Interventions (4 Programs): Four Programs utilized included DC perception and sub-perception; DR perception and subperception based programming
Period: Overall Study
Arm/Group | Subjects Received All Interventions (4 Programs)
Started | 2
DC Perception | 2
DR Perception | 2
DR Subperception | 2
DC Subperception | 1
Completed | 1
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Subjects Received 4 Interventions (4 Programs): Four Programs utilized included DC perception and sub-perception; DR perception and subperception based programming
Arm/Group | Subjects Received 4 Interventions (4 Programs)
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 59 [47 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity
Description: Change in pain intensity from Baseline to end of each Period (knee/foot).
  Pain scores are measured on a scale of 0 - 10 where 0 is no pain and 10 is maximum pain possible.
Time Frame: up to 6 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Dorsal Column (DC) Perception | Dorsal Root (DR) Perception | Dorsal Root (DR) Sub-perception | Dorsal Column (DC) Sub-perception
Number analyzed (Participants) | 2 | 2 | 2 | 1
units on a scale | 5 [4 to 6] | 4.5 [2 to 7] | 4.5 [2 to 7] | 1 [1 to 1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected and reported up to end of crossover phase (approximately 18 weeks)
Arm/Group | Dorsal Column (DC) Perception | Dorsal Root (DR) Perception | Dorsal Column (DC) Sub-perception | Dorsal Root (DR) Sub-perception
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/1 | 1/2
Other Adverse Events (participants affected / at risk) | 0/2 | 1/2 | 1/1 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dorsal Column (DC) Perception (N=2) | Dorsal Root (DR) Perception (N=2) | Dorsal Column (DC) Sub-perception (N=1) | Dorsal Root (DR) Sub-perception (N=2)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dorsal Column (DC) Perception (N=2) | Dorsal Root (DR) Perception (N=2) | Dorsal Column (DC) Sub-perception (N=1) | Dorsal Root (DR) Sub-perception (N=2)
Fasciculation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
No bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/46/NCT04073446/Prot_SAP_004.pdf